CLINICAL TRIAL: NCT05071131
Title: Investigating the Effect of Inulin on Gut Microbiota and Gut Barrier in Advanced Chronic Kidney Disease - a Randomised, Placebo-controlled Trial
Brief Title: Effect of Inulin on Gut Microbiota and Gut Barrier in Chronic Kidney Disease
Acronym: RESTORE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Till Schütte, Principle Investigator, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: RESTORE
Record Dates: First submitted 2021-09-16; First posted 2021-10-08 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Chronic Kidney Disease 5D
Keywords: Hemodialysis; Fiber; Zonulin; Short chain fatty acids; Dietary analysis
MeSH Terms: interventions — Inulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inulin (Active Comparator): 15 grams inulin per day for 7 days, followed by 30 grams inulin per day for 28 days
  Interventions: Dietary Supplement: Inulin
- Placebo (Placebo Comparator): 15 grams maltodextrin per day for 7 days, followed by 30 grams maltodextrin per day for 28 days
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Inulin — 1 sachet à 15 grams daily for 7 days, followed by 2 sachets à 15 grams daily for 28 days
  Arms: Inulin
Dietary Supplement: Placebo — 1 sachet à 15 grams daily for 7 days, followed by 2 sachets à 15 grams daily for 28 days
  Arms: Placebo

SUMMARY:
An adequate fiber intake is crucial for a well-balanced diet and reduces the risk of chronic diseases. However, nutritional recommendations for chronic kidney disease patients lead to an insufficient fiber intake with possible maladaptive effects on the gut microbiome. Therefore, we want to study the effects of a 35-day inulin supplementation on the gut microbiome, gut barrier function, bacterial metabolites and immune cell states in chronic kidney disease patients.

ELIGIBILITY:
Inclusion Criteria:

* Men and women in a ratio of 1:1
* Age 18-75 years
* Body mass index 25.0 - 39.9 kg/m^2
* End-stage kidney disease, which has been treated regularly with hemodialysis for at least 3 months

Exclusion Criteria:

* Malignant diseases
* Recent or current hospitalization
* Postoperative phase
* Acute infections
* Malnutrition
* Antibiotic treatment within the last 4 weeks
* Regular intake of probiotics and/or prebiotics
* Change of body weight of more than 2 kg in the month prior to study entry
* Known drug or alcohol abuse

Changes applied in July 2022 according to amendment no. 1:

* Two inclusion criteria were changed to improve recruitment

  * Age range was changed from 18-70 to 18-75 years
  * BMI range was changed from 18.5 - 34.9 to 25.0 - 39.9 kg/m^2
* The intervention scheme was adapted to increase patient adherence

  * A 7-day adaption phase with half of the dose (15 grams per day) at the start of the intervention was introduced, changing treatment duration from 28 to 35 days

Changes applied in January 2024 according to amendment no. 2:

* One inclusion criteria was changed to improve recruitment

  * BMI range was changed from 25 - 39,9 to 18,5 - 39,9 kg/m²
* Last visit was brought foward by 4 weeks.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Plasma concentration of Zonulin-1 | After 35 days compared to placebo
  Measured by ELISA [ng/ml]

SECONDARY OUTCOMES:
Plasma concentration of soluble CD14 | After 35 days compared to placebo
  Measured by ELISA [ng/ml]
Short-chain fatty acid-associated bacterial gene expression | After 35 days compared to placebo and adjusted for baseline
  Measured by quantitative PCR
Short-chain fatty acid-associated gene expression in immune cells | After 35 days compared to placebo
  Measured by quantitative PCR
Indole-associated bacterial gene expression | After 35 days compared to placebo
  Measured by quantitative PCR
Indole-associated gene expression in immune cells | After 35 days compared to placebo
  Measured by quantitative PCR
Fecal metabolome | After 35 days compared to placebo and adjusted for baseline
  Measured by mass spectrometry
Serum metabolome | After 35 days compared to placebo
  Measured by mass spectrometry
Serum concentration of Trimethylamine-N-Oxide (TMAO) | After 35 days compared to placebo
  Measured by LC-MS [µM]
Fecal microbiome taxonomy | After 35 days compared to placebo
  Measured by 16S amplicon sequencing
Activation potential of aryl hydrocarbon receptor (AhR) in serum | After 35 days compared to placebo and adjusted for baseline
  Measured by cell-based luciferase reporter assay (delta luminescence)
Frequency of circulating T-cell subtypes | After 35 days compared to placebo
  Measured by flow cytometry (%)
Office systolic blood pressure | After 35 days compared to placebo
  Mean of five consecutive blood pressure measurements (mmHg)
Office diastolic blood pressure | After 35 days compared to placebo
  Mean of five consecutive blood pressure measurements (mmHg)
Plasma concentration of IL-1 | After 35 days compared to placebo
  Measured by ELISA [pg/ml]
Plasma concentration of IL-6 | After 35 days compared to placebo
  Measured by ELISA [pg/ml]
Plasma concentration of TNF-alpha | After 35 days compared to placebo
  Measured by ELISA [pg/ml]
Creatinine | After 35 days compared to placebo
  Creatine serum concentration
Cystatin c | After 35 days compared to placebo
  Cystatin c serum concentration
Creatinine / cystatin c ratio | After 35 days compared to placebo
  Measured in serum

CONTACTS AND LOCATIONS:
Overall Officials: Anja Mähler, PhD, Principal Investigator — Charite University, Berlin, Germany; Nicola Wilck, MD, Principal Investigator — Charite University, Berlin, Germany; Victoria McParland, PhD, Principal Investigator — Charite University, Berlin, Germany; Johannes Holle, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Experimental and Clinical Research Center, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results of reported articles (text, tables, figures, supplemental data) will be shared after deidentification.
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal.